CLINICAL TRIAL: NCT05795413
Title: Patient Quality of Recovery From Mastectomy With and Without PECS Block With Liposomal Bupivacaine
Brief Title: Quality of Recovery From Mastectomy With and Without PECS Blocks
Status: Active, not recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Katharine Yao, MD, Chief, Division of Surgical Oncology Vice Chair, Research and Development, Endeavor Health
Other Study IDs: EH22-492
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Post Operative Pain; Quality of Recovery After Mastectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PECS Block with Liposomal Bupivacaine: The patients in this cohort will undergo a PECS block with Liposomal Bupivacaine before their mastectomy. Patients will receive Liposomal Bupivacaine in combination with 0.25% Bupivacaine in a 1:1 mixture for the purpose of post-operative pain control.
  Interventions: Procedure: Mastectomy with PECS blocks; Drug: Liposomal bupivacaine
- No PECS block: The patients in cohort will not undergo a PECS block. Pain will be controlled in the usual fashion with IV and oral medications.

INTERVENTIONS:
Procedure: Mastectomy with PECS blocks — Approximately half of patients recruited will receive a PECS block with Liposomal bupivacaine and half will not receive a block.
  Groups: PECS Block with Liposomal Bupivacaine
Drug: Liposomal bupivacaine — All of the PECS blocks performed at this institution have liposomal lupivacaine as the anesthetic. Investigators will examine quality of recovery and pain control in patients who receive a PECS block versus those who do not receive one.
  Groups: PECS Block with Liposomal Bupivacaine

SUMMARY:
This is a prospective observational study. Investigators want to understand post-operative recovery for patients undergoing mastectomy at NorthShore University HealthSystem. Some of these patients receive PECS blocks with Liposomal Bupivacaine and some do not receive a block. Investigators want to know whether patients who receive a block have better post operative recovery and pain control than patients who do not receive one. Investigators also want to understand whether PECS blocks with Liposomal Bupivacaine improves quality of recovery at 72 hours post operatively.

DETAILED DESCRIPTION:
Investigators plan to approach and consent 800 patients undergoing mastectomy, 400 with PECS blocks and 400 without. Investigators will assess their quality of recovery using the QoR 15 survey at 72 hours post operatively. In addition, investigators will also record VAS scores immediately postoperatively and at 24, 48, and 72 hours postoperatively. The study team will also calculate the total morphine equivalents (MMEs) required for each patient after 72 hours.

ELIGIBILITY:
Inclusion Criteria:

Must be female Must be >18 years old and < 90 years old Must be able to consent in English or Spanish May or may not have breast cancer (prophylactic mastectomy) Must be undergoing unilateral or bilateral mastectomy of any type May choose to proceed with or without breast reconstruction

Exclusion Criteria:

Allergy to all narcotic or local anesthetic medications Intake of any chronic opioids or pain medications preoperatively for a chronic condition or chronic use.

Subjects who received PECS blocks but whose block failed or is deemed not effective by an anesthesia provider as indicated by postoperative evaluation exam.

Vulnerable subjects (children, prisoners, pregnant women)

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females having mastectomy either for cancer diagnosis or prophylactic.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 15 Survey | 72 hours post operatively
  Patients will complete the quality of recovery 15 survey 72 hours after surgery. This is a scale from 0 to 150. A score of 150 indicates better post operative recovery.

SECONDARY OUTCOMES:
Visual analog scale | Immediately post operatively
  This is a pain scale from zero to ten. A score of 10 indicates worse pain.
Visual analog scale | 24 hours post operatively
  This is a pain scale from zero to ten. A score of 10 indicates worse pain.
Visual analog scale | 48 hours post operatively
  This is a pain scale from zero to ten. A score of 10 indicates worse pain.
Visual analog scale | 72 hours post operatively
  This is a pain scale from zero to ten. A score of 10 indicates worse pain.
Morphine milligram equivalents | Immediately post operatively
  We will record the amount of pain medication each patient takes after surgery. A higher morphine milligram equivalent indicates a higher amount of opioid medication used.
Morphine milligram equivalents | 24 hours post operatively
  We will record the amount of pain medication each patient takes after surgery. A higher morphine milligram equivalent indicates a higher amount of opioid medication used.
Morphine milligram equivalents | 48 hours post operatively
  We will record the amount of pain medication each patient takes after surgery. A higher morphine milligram equivalent indicates a higher amount of opioid medication used.
Morphine milligram equivalents | 72 hours post operatively
  We will record the amount of pain medication each patient takes after surgery. A higher morphine milligram equivalent indicates a higher amount of opioid medication used.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Yao, M.D., Principal Investigator — Endeavor Health
Locations (1):
- Evanston Hospital, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No